CLINICAL TRIAL: NCT02540694
Title: Endobronchial vs. Esophageal Ultrasound for Diagnosing Sarcoidosis: A Randomized Clinical Trial; - A Standard vs. - ProCore Needle Comparison -
Brief Title: EBUS vs EUS-B for Diagnosing Sarcoidosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Cook Medical (Unknown)
Responsible Party: Principal Investigator, L.M.M. Crombag, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL51598.018.15
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Sarcoidosis; Endosonography
MeSH Terms: conditions — Sarcoidosis | interventions — Endosonography

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- EBUS-TBNA using 22G needle (Active Comparator): EBUS-TBNA using 22G needle (transbronchial route)
  Interventions: Device: Endosonography
- EBUS-TBNA using 25G ProCore needle (Active Comparator): EBUS-TBNA using 25G ProCore needle (transbronchial route)
  Interventions: Device: Endosonography
- EUS-B-FNA using 22G needle (Active Comparator): EUS-B-FNA using 22G needle (transoesophageal route)
  Interventions: Device: Endosonography
- EUS-B-FNA using 25G ProCOre needle (Active Comparator): EUS-B-FNA using 25G ProCOre needle (transoesophageal route)
  Interventions: Device: Endosonography

INTERVENTIONS:
Device: Endosonography
  Other Names: EBUS; EUS-B

SUMMARY:
Rationale:

Endosonography with mediastinal/ hilar nodal sampling is the test of choice to diagnose sarcoidosis stage I and II - in case tissue verification of noncaseating granulomas is indicated. However, the optimal endosonographic approach (endobronchial or transoesophageal) for mediastinal nodal sampling is under discussion.

Secondly, which needle size or type provides optimal tissue sample quality for granuloma detection is unknown. The novel 25 Gauge (G) beveled ProCore needle, allows tissue acquisition of small core biopsies in addition to cytological aspirates.

Hypotheses:

1. Esophageal ultrasound guided (EUS-B) sampling of intrathoracic lymph nodes has a 14% higher granuloma detection rate compared to endobronchial ultrasound (EBUS) guided nodal sampling in patients with suspected sarcoidosis stage I/II.
2. 25G ProCore needles provide superior sample quality compared to conventional 22G needles in patients with suspected sarcoidosis stage I/II.

Study design:

Investigator initiated, randomized clinical trial. Setting: International, multicenter (university and general hospitals)

Study population:

Consecutive patients with a clinical and radiologic suspicion of sarcoidosis stage I or II and an indication for tissue verification of non-caseating granulomas are eligible for inclusion.

Intervention:

EBUS vs EUS-B, simultaneously comparing the standard vs novel ProCore needles.

Main study endpoints:

1. The granuloma detection rate of endobronchial (EBUS) guided sampling of intrathoracic lymph nodes compared to esophageal (EUS-B using the EBUS scope) guided sampling in patients with suspected sarcoidosis stage I/II.
2. Sample quality of conventional 22G vs. 25G ProCore needles in patients with suspected sarcoidosis stage I/II.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiologic suspicion of sarcoidosis stage I (mediastinal or hilar lymphadenopathy) or stage II (lymphadenopathy and interparenchymal abnormalities)
* Indication for tissue verification of noncaseating granuloma's
* Provision of a written informed consent

Exclusion Criteria:

* Life expectancy of less than 6 months
* Obvious organ involvement of sarcoidosis with the possibility to confirm granulomas with a minimally invasive diagnostic procedure (eg skin lesion or superficial lymph node)
* Positive acid-fast bacilli sputum test
* Contra-indication for endosonography
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-11 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The granuloma detection rate of endobronchial (EBUS) guided sampling of intrathoracic lymph nodes compared to esophageal (EUS-B using the EBUS scope) guided sampling in patients with suspected sarcoidosis stage I/II. | 2 weeks after the endosonography procedure.
Sample quality of conventional 22G vs. 25G ProCore needles in patients with suspected sarcoidosis stage I/II. | 9 months after inclusion of last patient.
  The sample quality will be assessed by two independent reference pathologists. The performance of each needle (25 ProCore / standard 22 G) will be scored on five items (the modified Mair score).

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, Prof, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Amsterdam, Netherlands

REFERENCES:
- [Derived] Crombag LMM, Mooij-Kalverda K, Szlubowski A, Gnass M, Tournoy KG, Sun J, Oki M, Ninaber MK, Steinfort DP, Jennings BR, Liberman M, Bilaceroglu S, Bonta PI, Korevaar DA, Trisolini R, Annema JT. EBUS versus EUS-B for diagnosing sarcoidosis: The International Sarcoidosis Assessment (ISA) randomized clinical trial. Respirology. 2022 Feb;27(2):152-160. doi: 10.1111/resp.14182. Epub 2021 Nov 17. PMID 34792268